CLINICAL TRIAL: NCT02049632
Title: Survival and Axillary Relapse in Breast Cancer Patients With Sentinel Node Micrometastases Who Have Not Undergone Completion Axillary Clearance - a National Cohort Study
Brief Title: Sentinel Node Biopsy in Breast Cancner: Omission of Axillary Clearance After Micrometastasis
Acronym: SENOMIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Centrallasarettet Västerås (Other); Uppsala University (Other)
Responsible Party: Principal Investigator, Jana de Boniface, MD, PhD, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SENOMIC
Record Dates: First submitted 2014-01-24; First posted 2014-01-30 (Estimated); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Sentinel Node Biopsy; Micrometastasis; Axillary lymph node dissection
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Micrometastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omission of axillary clearance (Experimental): No axillary lymph node dissection after sentinel node biopsy and sentinel node micrometastases
  Interventions: Procedure: Omission of axillary clearance

INTERVENTIONS:
Procedure: Omission of axillary clearance

SUMMARY:
Sentinel node (SN) biopsy in breast cancer has been demonstrated to be a reliable method, and several follow-up studies have shown that it is safe to refrain from completion axillary clearance (axillary lymph node dissection, ALND) in SN-negative patients. SN biopsy alone results in significantly less arm discomfort following the operation.

However, as a surprisingly low frequency of axillary relapse has been observed in patients without any axillary intervention (neither SN biopsy nor axillary clearance), or without completion ALND after a positive SN biopsy, the importance of ALND is being questioned, even for patients with SN metastases. A large, randomized study (ISBCG23-1) was not able to show any differences in 5-year disease-free survival between patients with SN micrometastases who had undergone ALND and those who had not.

This Swedish multicenter study will include patients with SN micrometastases. These women will not undergo ALND but will be registered in a study cohort. The patients will otherwise be treated in accordance with the national guidelines and will be clinically followed every year for five years, after 10 years and finally after 15 years. Hypothesis: To refrain from axillary clearance in breast cancer patients with sentinel node micrometastases does not impair survival.

DETAILED DESCRIPTION:
From April 2017 onwards, only patients operated by mastectomy or those receiving neoadjuvant therapy and having a sentinel node biopsy before its initiation may be recruited into SENOMIC. The inclusion target has been met for those patients operated by breast-conserving therapy, and from now on, these patients will not be included in SENOMIC anymore. Recruitment of the above-mentioned patient selection will continue until 452 patients operated by mastectomy have been enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically node-negative, invasive breast cancer ≤ 5 cm (T1-T2)
* Histopathology results demonstrate SN micrometastases.
* Patients who undergo mastectomy (protocol change from April 2017 onwards)
* The patient must have given verbal and written consent.

Exclusion Criteria:

* Preoperatively diagnosed lymph node metastases.
* Sentinel node metastases > 2 mm.
* Metastases beyond the ipsilateral axillary lymph nodes at the time of surgery.
* History of previous breast cancer.
* Pregnancy.
* Bilateral breast cancer where any of the other exclusion criteria applies to either side.
* Medical contraindication for systemic adjuvant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 805 (Actual)
Dates: Start 2013-12; Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | Five years

SECONDARY OUTCOMES:
Axillary recurrence rate | Five years

OTHER OUTCOMES:
Breast cancer-specific survival | Five years
Overall survival | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Jana M de Boniface, MD, PhD, Principal Investigator — Karolinska Institutet; Jan Frisell, Professor, Principal Investigator — Karolinska Institutet; Leif Bergkvist, Professor, Principal Investigator — Uppsala University; Yvette Andersson, MD, PhD, Principal Investigator — Västmanlands Hospital
Locations (22):
- Sweden (22):
  - Sahlgrenska University Hospital, Gothenburg
  - Helsingborgs Hospital, Helsingborg
  - Kalmar Hospital, Kalmar
  - Karlskrona Hospital, Karlskrona
  - Kristianstad Hospital, Kristianstad
  - Lidköping Hospital, Lidköping
  - Linköping University Hospital, Linköping
  - Lund and Malmö University Hospital, Lund
  - Örebro University Hospital, Örebro
  - Skövde Hospital, Skövde
  - Karolinska University Hospital, Stockholm
  - Capio St Görans Hospital, Stockholm
  - Danderyds Hospital AB, Stockholm
  - Southern General Hospital, Stockholm
  - Sundsvall Hospital, Sundsvall
  - Uddevalla Hospital, Uddevalla
  - Umeå University Hospital, Umeå
  - Akademiska Universitetssjukhuset, Uppsala
  - Varberg Hospital, Varberg
  - Växjö Hospital, Vaxjo
  - Västmanlands Hospital, Västerås
  - Västervik Hospital, Västervik